CLINICAL TRIAL: NCT06966466
Title: Effects of Deep Touch Pressure on Emergence Agitation in Pediatric Patients Undergoing Tonsillectomy and Adenoidectomy: A Prospective Randomized Controlled Study
Brief Title: Effects of Deep Touch Pressure on Emergence Agitation in Pediatric Patients
Acronym: HUGGY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2503-017-1620
Record Dates: First submitted 2025-05-09; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Deep Touch Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DTP group (Experimental)
  Interventions: Device: HuGgy Compression vest
- Control group (No Intervention)

INTERVENTIONS:
Device: HuGgy Compression vest — This intervention involves the use of a HUGgy compression vest, a wearable device that provides deep touch pressure (DTP) to pediatric patients undergoing tonsillectomy and adenoidectomy under general anesthesia. The vest is worn by patients immediately after surgery, and pressure is applied to provide calming sensory input. The pressure level is adjusted based on the manufacturer's guidelines, providing a gentle, even compression to reduce emergence agitation (EA) during the recovery period.
  Arms: DTP group

SUMMARY:
The goal of this clinical trial is to determine if deep touch pressure (DTP) can reduce emergence agitation (EA) in pediatric patients aged 3 to 10 years undergoing tonsillectomy and adenoidectomy under general anesthesia. The main questions it aims to answer are:

Does deep touch pressure (DTP) using a compression vest reduce the incidence of emergence agitation (EA) in the recovery room?

Does DTP reduce the severity of EA, as measured by the Pediatric Assessment of Emergence Delirium (PAED) scale?

Researchers will compare:

Intervention Group: Pediatric patients who receive DTP using the HUGgy compression vest during the recovery period.

Control Group: Pediatric patients who receive standard postoperative care without DTP.

Participants will:

Be randomly assigned to either the intervention group (DTP) or the control group.

Undergo standard general anesthesia for tonsillectomy and adenoidectomy.

Wear the HUGgy compression vest if assigned to the intervention group.

Be monitored for emergence agitation using the PAED scale and FLACC pain scale in the recovery room.

Receive rescue medication (nalbuphine) if severe EA occurs.

This study will help determine if DTP can be used as a safe and effective non-pharmacological method to reduce emergence agitation in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 3 to 10 years scheduled for tonsillectomy and adenoidectomy under general anesthesia.

Exclusion Criteria:

* Emergency surgery.
* Known neurological disorders (e.g., epilepsy, cerebral palsy).
* Skin disorders or injuries on the chest or upper body that prevent safe use of the compression vest (HUGgy).
* History of severe psychiatric disorders (e.g., autism spectrum disorder, severe anxiety disorder).
* History of severe allergic reactions to anesthesia.
* Any condition that, in the investigator's judgment, makes the patient unsuitable for the study.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Emergence Agitation in Post-anesthesia care unit | Within 30 minutes of recovery room admission.
  The incidence of emergence agitation (EA) is defined as a PAED (Pediatric Assessment of Emergence Delirium) scale score greater than 10 within the first 30 minutes after admission to the post-anesthesia care unit

SECONDARY OUTCOMES:
Maximum PAED Scale Score in Post-Anesthesia Care Unit | From PACU admission to discharge (up to 1 hour)
  From PACU admission to discharge (up to 1 hour).
Incidence of Severe Emergence Agitation (EA) in PACU | From PACU admission to discharge (up to 1 hour)
Maximum FLACC Pain Score in PACU | From PACU admission to discharge (up to 1 hour)
Duration of PACU Stay | From PACU admission to discharge (up to 1 hour)
Use of Rescue Medication in PACU | From PACU admission to discharge (up to 1 hour)
Compliance with Deep Touch Pressure (DTP) Intervention | From PACU admission to discharge (up to 1 hour)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Children's Hospital, Seoul, Seoul, South Korea